CLINICAL TRIAL: NCT06942325
Title: Performance and Effectiveness of a Self-fitting Over-the-counter Hearing Aid in Adults With Perceived Mild-Moderate Hearing Loss: A Three Phased Approach
Brief Title: Performance and Effectiveness of a Self-fitting Over-the-counter Hearing Aid
Acronym: Lexie
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn before enrollment for administrative reasons.
Sponsor: HearX SA (Industry)
Responsible Party: Sponsor
Organization: hearX Group (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Lexie
Record Dates: First submitted 2025-03-11; First posted 2025-04-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hearing Loss; Hearing Impairment
Keywords: hearing loss; over-the-counter hearing aid; self-fitting hearing aid; prescription hearing aid
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OTC SF Group (Experimental): Participants in this group will field trial a self-fitting over-the-counter (OTC SF) hearing aid. Each participant will independently set up and adjust their device without any professional assistance, following standard self-fitting procedures. They will receive only the manufacturer-provided instructional materials, including the user manual and quick start guide, as would be typical for real-world OTC hearing aid use. This process reflects the intended consumer-directed experience for OTC hearing aids.
  Interventions: Device: OTC self-fitting hearing aid
- Prescription Group (Active Comparator): Participants in this group will use a professionally fitted prescription hearing aid. A licensed audiologist will conduct a comprehensive hearing evaluation, followed by device selection (receiver wires and domes), programming, and individualized fitting based on best practice protocols. The fitting will be fine-tuned using real-ear measurements (REM) to ensure optimal amplification settings tailored to each participant's hearing profile. Additionally, participants will receive professional counseling on device use, care, and expectations, reflecting the standard clinical hearing aid fitting process.
  Interventions: Device: Prescription hearing aid

INTERVENTIONS:
Device: OTC self-fitting hearing aid — OTC hearing aid to be compared to prescription hearing aid
  Other Names: OTC hearing aid
  Arms: OTC SF Group
Device: Prescription hearing aid — Prescription hearing aid used as active comparator to the OTC self-fitting hearing aid
  Arms: Prescription Group

SUMMARY:
Hearing loss significantly affects quality of life, with sensorineural hearing loss being the most common type among adults. Hearing aids are a proven intervention, yet barriers like access and affordability limit their adoption, even in high-income countries with developed audiological services . Traditionally, hearing aids required professional consultations, restricting access. However, in 2022, the U.S. FDA approved over-the-counter (OTC) hearing aids, including self-fitting devices, to improve accessibility. Recent clinical trials suggest that OTC hearing aids can deliver similar benefits to professionally fitted ones in speech recognition and self-reported outcomes.

Critiques of these studies have focused on using the same device model for both groups rather than comparing it to established prescription hearing aids. To address this, the current study employs a phased approach. Phase 1 validates an in-situ hearing test against a standard audiometer, Phase 2 assesses user experience, and Phase 3 involves a randomized control trial comparing a self-fitting OTC hearing aid with a professionally fitted prescription device. The hypothesis is that both devices offer equivalent benefits.

This research is novel as no previous studies have directly compared self-fitting OTC and commercially available prescription hearing aids. This study will compare the effectiveness of an OTC self-fitting hearing aid against a prescription device using a crossover randomized control trial.

DETAILED DESCRIPTION:
Hearing loss is a prevalent condition affecting a significant portion of the global population, leading to challenges in communication, social interactions, and overall quality of life. Recent data indicates that over 1.5 billion individuals worldwide experience some degree of hearing loss, with 430 million facing disabling hearing impairments. For adults with sensorineural hearing loss, hearing aids are the primary intervention to enhance auditory function. Conventionally, obtaining hearing aids involves comprehensive diagnostic assessments, device selection, and personalized fitting conducted by hearing care professionals. While this method ensures tailored care, it can also pose accessibility challenges, including financial constraints, limited availability of trained professionals, and social stigma associated with hearing aid use. These barriers contribute to the limited adoption and underutilization of hearing aids, even in regions with adequate audiological services.

To address these accessibility issues, over-the-counter (OTC) hearing aids have been introduced as a viable alternative. This model empowers individuals with perceived mild to moderate hearing loss to independently select and fit hearing aids without the necessity of professional evaluations. The U.S. Food and Drug Administration (FDA) established regulations for OTC hearing aids, which took effect on October 17, 2022. These regulations aim to increase accessibility and affordability of hearing care solutions. The introduction of OTC hearing aids represents a shift towards consumer hearing care. By allowing individuals to manage their hearing needs independently, OTC hearing aids have the potential to reduce barriers associated with traditional hearing aid procurement, such as high costs and limited access to audiologists. This newer model of care aligns with a broader public health goal to enhance the availability of hearing aids.

Recent clinical trials have indicated that over-the-counter (OTC) hearing aids can provide benefits comparable to those of professionally fitted devices, particularly in the areas of user-reported satisfaction. For instance, a randomized clinical trial compared the effectiveness of a self-fitting OTC hearing aid with remote support to that of an audiologist-fitted device. The study found that self-reported outcomes and speech recognition in noise benefits were noninferior in the self-fitting group compared to the audiologist-fitted group. Despite these promising findings, critiques have emerged regarding the methodologies of this and other similar studies. A primary concern is that many studies utilize the same device model for both the OTC and professionally fitted groups, rather than comparing OTC devices to established prescription hearing aids. This approach may limit the generalizability of the results, as it does not account for the variability in performance across different hearing aid models. Therefore, there is a need for studies that compare self-fitting OTC hearing aids directly with prescription devices to provide a more comprehensive understanding of their relative effectiveness. The aim of this randomized controlled trial is to compare the effectiveness of a self-fitting OTC hearing aid to a prescription hearing aid. This trial forms a part of a larger validation study, that includes two other phases (validating an in-situ hearing test and usability assessment of the self-fitting OTC hearing aid). However, we describe here only the effectiveness trial (Phase 3). The hypothesis is that the self-fitting OTC hearing aid will provide non-inferior benefits compared to the professionally fitted prescription hearing aid in terms of user-reported outcomes and speech recognition in noise. Several other exploratory measures will also be evaluated through the course of the trial.

ELIGIBILITY:
Inclusion criteria:

* Participant must be 18 years or older.
* The outer ear must be free from excessive cerumen, outer or middle ear disease (determined through otoscopic examination of the ear)
* The participant must have bilateral self-perceived mild-moderate hearing loss.
* Baseline pure tone evaluations should fall within a 4-frequency PTA (0.5, 1.0, 2.0, 4.0 kHz) of 65 dB HL or less.
* The participant must have an adequate level of English proficiency as measured objectively using an English proficiency test (EF SET).
* The participant must have Type A or As or Ad tympanogram as measured by tympanometry.
* Must be in possession of a smartphone compatible with the Lexie App (minimum iOS 13 or Android OS 10), preferably within equal distributio

Exclusion Criteria:

* Younger than 18 years
* Presents with severe or greater hearing loss in either ear
* Presents with an outer or middle ear abnormality

Have any of the following as per FDA (21 CFR 801.420) reg-flag conditions as contraindications to OTC hearing aid use :

(i) Visible congenital or traumatic deformity of the ear preventing insertion of the receiver wire and dome into the ear.

(ii) History of sudden active drainage (i.e. blood or pus) from the ear within the previous 6 months.

(iii) Painful or uncomfortable feeling in your ear (iv) Visible evidence of significant cerumen accumulation or a foreign body in the ear canal.

(v) History of sudden or rapidly progressive hearing loss within the previous 6 months.

(vi) Acute or chronic dizziness. (vii) Unilateral hearing loss. (viii) Fluctuating hearing loss (ix) Unilateral tinnitus

* Low English proficiency - <51% of EF-SET
* No access or in possession of a smartphone, compatible with the Lexie App (minimum iOS 13 or Android OS 10)

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Abbreviated Profile of Hearing Aid Benefit (APHAB) | Baseline, three weeks and six weeks
  The APHAB will be the primary effectiveness endpoint measure for the trial. It is a standardised questionnaire used to assess the effectiveness of hearing aids. It measures the user's perceived hearing difficulties in various everyday situations both with and without their hearing aids, across four subscales: ease of communication, reverberation, background noise, and aversiveness of sounds. The results help to quantify the benefits and limitations of hearing aid use from the user's perspective. The APHAB global score is calculated by averaging the scores across three specific subscales of the APHAB: Ease of Communication, Reverberation, and Background Noise and will serve as the primary effectiveness outcome variable for the study phase. Patients report the percentage of time they experience difficulty in each situation (1% - 99%), with and without hearing aids. Benefit is calculated by comparing the unaided and aided scores, with higher benefit scores indicating better outcomes.

SECONDARY OUTCOMES:
International Outcome Inventory for Hearing Aids (IOI-HA) | Three weeks and six weeks
  The IOI-HA is a standardised questionnaire designed to evaluate the overall effectiveness and user satisfaction with hearing aids. It consists of seven items that assess key aspects such as daily use, benefit, residual activity limitations, satisfaction, residual participation restrictions, impact on others, and quality of life. The scale is ordinal in nature, but a total score can be calculated as the sum of all seven items. Each item is rated on a 5-point scale, with higher scores indicating more favorable outcomes. The total score ranges from 7 to 35, with higher scores reflecting greater benefit and satisfaction from hearing aid use.
Quick Speech in Noise Test (QuickSIN) | Baseline, three weeks and six weeks
  The QuickSIN is a clinically used assessment tool designed to evaluate an individual's ability to understand speech in noisy environments by presenting speech in multi-talker babble noise. During the test, six sentences-each containing five key words-are presented with four-talker babble noise. The speech level decreases in 5 dB steps from a signal-to-noise ratio (SNR) of 25 dB to 0 dB. Patients repeat each sentence, and clinicians score one point for each correctly repeated key word, totaling up to 30 points per list. The SNR loss is calculated by subtracting the total correct words from 25.5. Lower SNR loss values indicate better speech understanding in noisy environments. Three lists will be completed at each assessment point, and the average SNR of the three lists will be used for the final calculation.
Real ear aided response (REAR) | Three weeks and six weeks
  REAR is a measure used to evaluate the sound level at the eardrum when a hearing aid is worn and active. It captures how the hearing aid amplifies sound across different frequencies directly in the user's ear canal.
  In relation to NAL-NL2 targets, REAR is used to verify that the hearing aid's amplification matches the prescribed targets set by the NAL-NL2 fitting formula. NAL-NL2 is a widely used prescriptive method for fitting hearing aids, aiming to optimise speech intelligibility while maintaining comfort. During a fitting, the audiologist measures the REAR and compares it to the NAL-NL2 targets to ensure that the hearing aid is providing the appropriate gain for the user's specific hearing loss, ensuring optimal hearing aid performance and user satisfaction. We will determine how far the REAR is from NAL-NL2 prescriptive target in decibel sound pressure level [dB SPL] at 0.5, 1,2 and 4 kHz. A lower number in dB SPL (NAL-NL2 target - REAR) suggests closer alignment to target.

OTHER OUTCOMES:
Revised Hearing Handicap Inventory - Screening (RHHI-S) | Baseline, three weeks and six weeks
  The RHHI-S is a tool designed to quickly assess the perceived impact of hearing loss on an individual's social and emotional well-being. It is often used in clinical and screening settings to identify individuals who may be experiencing difficulties due to hearing loss and who might benefit from further audiological evaluation or intervention. It consists of 10 items, with possible scores ranging from 0 to 40. Each item is answered with "Yes" (4 points), "Sometimes" (2 points), or "No" (0 points). Higher scores indicate a greater perceived hearing handicap. A score of 10 or higher suggests a significant hearing handicap, warranting further audiological evaluation.
Hearing aid skills and knowledge inventory-clinician (HASKI-Clin) | Three weeks and six weeks
  The HASKI-clin is a tool used by clinicians to assess a hearing aid user's ability to manage and maintain their devices effectively. It evaluates key skills and knowledge areas, such as inserting and removing the hearing aids, changing batteries, adjusting volume, cleaning and maintaining the devices, and troubleshooting common issues. The HASKI-clin comprises 35 items focusing on skills necessary for daily hearing aid use, maintenance, and minor repairs. To calculate the competency percentage, the number of competent items are divided by the total applicable items and multiplied by 100. A higher percentage indicates greater competency, with 100% representing full proficiency. Each item is equally weighted, reflecting the diverse challenges individuals might face with different tasks.
Generalized Self Efficacy Scale (GSES) | Baseline
  The GSES is a 10-item questionnaire designed to assess an individual's overall belief in their ability to handle various challenging situations and achieve goals. Each of the 10 items is rated on a 4-point Likert scale and a total score is obtained by summing the responses across the 10 items, which can range from 10 - 40. A higher score indicates greater self-efficacy.
Digital Literacy 2-Question (DL-2Q) | Baseline
  The DL-2Q is a brief, validated tool consisting of two questions designed to assess an individual's proficiency and confidence in using mobile devices. The first question evaluates the user's skill level with a mobile device on a scale from 0 ("never used a mobile device") to 2 ("competent"), while the second question measures their confidence in using a mobile device, also on a scale from 0 ("not confident and usually need help") to 2 ("confident"). The DL-2Q was developed to specifically address the growing importance of digital literacy, particularly in older adults, in the context of mobile technology use. It provides a quick and effective way to gauge digital literacy, especially in populations participating in digital intervention studies.
Expected Consequences of Hearing Aid Ownership (ECHO) | Baseline
  The ECHO is a self-assessment tool designed to evaluate an individual's expectations regarding hearing aid use before they acquire one. It measures expectations across several domains, including positive effects (such as improved communication), service and cost (expectations about follow-up care and financial considerations), negative features (potential drawbacks of hearing aid use), and personal image (concerns about appearance and social stigma). Each of the 15 items is rated on a 7-point Likert scale and the responses are summed for total and subscale scores. The total score is the sum of all items scored, a higher score indicating more positive expectations).
Patient Global Impression of Change (PGI-C) | Three weeks and six weeks
  The PGI-C is a single-item self-report measure that assesses a patient's overall perception of improvement or decline in their condition over time. Patients rate their change on a 7-point scale ranging from "no change" to "a great deal better" or "a great deal worse." The PGI-C is commonly used in clinical trials to capture a subjective sense of treatment effectiveness from the patient's perspective, offering valuable insight into the perceived impact of interventions
Data logging | Three weeks and six weeks
  Data logging will be included to gain additional insights into the usage patterns of the self-fitted (SF) and audiologist-fitted (AF) hearing aids. Data logging refers to the automatic recording of specific metrics by the hearing aids during their use. These metrics can include a variety of factors, such as the total hours of use, average daily/ weekly hours of usage, and other user interactions with the device. Data will be logged according to daily hours of use.
Hearing aid perception questionnaire (self-developed) | Three weeks and six weeks
  Likert scale questions will be asked from participants to gain additional insights on their overall perception of the OTC self-fitting hearing aid features and experience with using the self-fit OTC and prescription hearing aid, following completion with each field trial. No particular scoring will be used. This questionnaire is to obtain descriptive perceptions of the two devices.

CONTACTS AND LOCATIONS:
Overall Officials: Karina C De Sousa, PhD, Principal Investigator — hearX Group

IPD SHARING:
Plan to Share IPD: No
The study is conducted under the South African Health Products Regulatory Authority (SAHPRA) and US Food and Drug Administration (FDA) Institutional regulations, which impose strict guidelines on the handling and sharing of medical device trial data. Furthermore, the data may contain proprietary or commercially sensitive information related to the device's performance. Sharing IPD could compromise intellectual property or competitive interests of the device manufacturer. While the raw IPD will not be shared, aggregate-level data, summary statistics, and study findings may be published and made available in peer-reviewed journals and reports.